CLINICAL TRIAL: NCT00079651
Title: Programming for Dementia: Maximizing Abilities
Brief Title: Montessori-Based Activities for Elderly Persons With Dementia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Menorah Park (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: R21MH063395 (NIH); R21MH063395 (NIH); DATR A4-GPS
Record Dates: First submitted 2004-03-10; First posted 2004-03-12 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Dementia
Keywords: Aged; Nursing Homes; Assisted Living Facilities
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Montessori-based dementia programming

SUMMARY:
This study will determine whether montessori-based activities can help older adults with dementia become more responsive to others.

DETAILED DESCRIPTION:
Studies have shown that Montessori-based activities, which focus on developing an individual's unique abilities, are effective in increasing engagement between nursing home residents with dementia and their caregivers. This study will determine whether the positive effects of Montessori-based programming can be replicated in adult day care, assisted living, and nursing homes. Results from this study will be used to create training materials to help staff in different settings implement the intervention within existing schedules, staffing, and programming routines.

This study will be conducted in two phases. During Phase I, participants with mild dementia will be trained to become small group leaders for Montessori-based activities. In Phase II, newly-trained participants will use their skills to assist others. Assessments will be made throughout the study. Participants' engagement with the environment and caregiver burden and satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia
* Living in or attending programs at participating sites

Exclusion Criteria:

* Medical conditions that would interfere with study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-12; Primary Completion 2005-04 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron J. Camp, PhD, Principal Investigator — Myers Research Institute
Locations (5):
- United States (5):
  - Mandel Adult Day Program, Beachwood, Ohio
  - Stone Gardens, Beachwood, Ohio
  - Eliza Bryant Village, Cleveland, Ohio
  - Jennings Center for Older Adults, Cleveland, Ohio
  - The Greens Adult Living Communities, Lyndhurst, Ohio

REFERENCES:
- See also: Click here to contact Myers Research Institute regarding this study — http://www.myersresearch.org